CLINICAL TRIAL: NCT04621266
Title: Effectiveness of a Home-based Peer Support Program for Chinese Mothers With Low Breastfeeding Self-efficacy to Increase the Exclusivity and Duration of Breastfeeding: a Randomized Controlled Trial
Brief Title: Home Based Peer Support Program for Mothers With Low Breastfeeding Self-efficacy
Acronym: BFPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BFPS1
Record Dates: First submitted 2020-10-29; First posted 2020-11-09 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2023-08

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Home-based peer support intervention (Experimental): Participants will receive intervention on top of standard usual care.
  Interventions: Behavioral: Online Home-based peer support
- Standard usual care (No Intervention): Participants will receive standard usual care.

INTERVENTIONS:
Behavioral: Online Home-based peer support — Online Home-based peer support will be provided to support participants' breastfeeding. There will be a minimum of 2 and maximum of 3 home visits between trained peer counsellors and participants. Each session will last approximately 30 minutes.
  Arms: Online Home-based peer support intervention

SUMMARY:
An online home-based breastfeeding peer support programme is proposed to support mothers who are giving birth to their first-born. This study aims to evaluate the effectiveness of this programme in improving breastfeeding practices among women with low breastfeeding self-efficacy. It is hypothesized that participants who received online home-based peer support will exclusively breastfeed for longer duration, have higher breastfeeding self-efficacy, and lower post-partum depression symptoms when compared to those receiving only standard care.

DETAILED DESCRIPTION:
Primiparous mothers who plan to breastfeed but did not go on to breastfeed often face high levels of emotional and psychological challenges in their transition to parenthood. This can adversely affect their breastfeeding experiences and general well-being, and is associated with stress, anxiety, and postnatal depression. While family psycho-education and other supportive group programmes are available in health services, they require face-to-face education sessions over a long interval, high engagement, and trusting relationships, and thus often result in low attendance and high drop outs.

Mothers have expressed the need for psychological support of peer counsellors, which would allow them to support each other. The first month postpartum is a critical period for sustaining exclusive breastfeeding and the time when mothers are at high risk of postpartum depression. For Chinese mothers in Hong Kong, however, they are often housebound during this period due to the tradition of "doing the month", and thus often find it difficult to attend support groups or seek help. In view of these challenges and the pandemic wave faced by primiparous mothers, they are reluctant with home visits, therefore an online delivery of the home-based peer support programme is proposed.

This randomized control trial adopts a two-arm design to examine the effectiveness of an online home-based peer support programme for women with low breastfeeding self-efficacy. It is hypothesized that those receiving the intervention, when compared to the controls, will have (1) longer period of exclusive breastfeeding, (2) higher postnatal breastfeeding self-efficacy, and (3) lower post-partum depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous mothers
* Intend to breastfeed
* Have low breastfeeding self-efficacy (between 14 to 32)
* Have singleton pregnancy and live birth
* Have term infant (37-42 weeks gestational)
* Cantonese speaking
* Hong Kong resident
* Have no serious medical or obstetrical complications

Exclusion Criteria:

* Infant is <37 week gestation
* Infant has Apgar score <8 at five minutes
* Infant has birthweight <2,500 grams
* Infant has any severe medical conditions or congenital malformations
* Infant is placed in the special care baby unit for more than 48 hours after birth
* Infant is placed in the neonatal intensive care unit at any time after birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kris YW Lok, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lok KYW, Choi MSL, Ko RWT, Chau PPH, Lam CCO, Chang YS, Bick D. Effectiveness of a home-based peer support programme for Chinese mothers with low breastfeeding self-efficacy to increase the exclusivity and duration of breastfeeding: study protocol of a randomised control trial. BMJ Open. 2024 Jul 23;14(7):e081897. doi: 10.1136/bmjopen-2023-081897. PMID 39043588

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Started | 224 | 218
Completed | 214 | 214
Not Completed | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care | Total
Number analyzed (Participants) | 224 | 218 | 442
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 224 | 218 | 442
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 218 | 442
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Infant Feeding Status: Exclusive Breastfeeding
Description: Number/ proportion of participants who practice exclusive breastfeeding at 1 months postpartum.
Time Frame: At 1 month postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 224 | 218
Participants | 46 | 39

2. Primary Outcome: Infant Feeding Status: Exclusive Breastfeeding
Description: Number/ proportion of participants who practiced exclusive breastfeeding at 2 month postpartum.
Time Frame: At 2 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 224 | 218
Participants | 54 | 38

3. Primary Outcome: Infant Feeding Status: Exclusive Breastfeeding
Description: Number/ proportion of participants that practice exclusive breastfeeding at 4 months postpartum.
Time Frame: At 4 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 224 | 218
Participants | 47 | 42

4. Primary Outcome: Infant Feeding Status: Exclusive Breastfeeding
Description: Number/ proportion of participants that practice exclusive breastfeeding at 6 months postpartum.
Time Frame: At 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 224 | 218
Participants | 37 | 29

5. Secondary Outcome: Women's Self-efficacy in Breastfeeding
Description: Breastfeeding Self-efficacy Scale Short Form (Hong Kong Chinese version) is used to measure maternal breastfeeding self-efficacy. The 14-item scale is on a 5-point Likert scale. Total score ranged from 14 to 70 with a higher score indicating higher breastfeeding confidence and self-efficacy. A cut-off score of 46 is applied after rounding up to the nearest integer.
Time Frame: At baseline, 2 months and 4 months postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 223 | 216
score on a scale | 45 (12.9) | 40.7 (11.3)

6. Secondary Outcome: Women's Self-efficacy in Breastfeeding at Baseline
Description: as for outcome 5
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 223 | 216
score on a scale | 37 (6.6) | 37 (6.6)

7. Secondary Outcome: Women's Self-efficacy in Breastfeeding at 2 Months Postpartum
Description: as for outcome 5
Time Frame: At 2 months postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 223 | 216
score on a scale | 40.6 (12.4) | 38.7 (6.6)

8. Secondary Outcome: Women's Self-efficacy in Breastfeeding at 4 Months Postpartum
Description: as for outcome 5
Time Frame: At 4 months postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 223 | 216
score on a scale | 45 (12.9) | 38.7 (6.6)

9. Secondary Outcome: Women's Postpartum Depression at Baseline
Description: The Chinese version of the Edinburgh Postnatal Depression Scale is used to measure the severity of postnatal depressive symptoms. It is a ten-item scale rated from 0 to 3. The total score could range from 0 to 30. In general, a higher score indicates more severe depressive symptoms.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 223 | 216
score on a scale | 8.2 (4.9) | 7.9 (4.4)

10. Secondary Outcome: Women's Postpartum Depression at 1 Month Postpartum
Description: as for outcome 9
Time Frame: At 1 month postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 223 | 216
score on a scale | 9.0 (4.5) | 8.8 (4.7)

11. Secondary Outcome: Women's Postpartum Depression at 2 Month Postpartum
Description: as for outcome 9
Time Frame: At 2 month postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
Number analyzed (Participants) | 223 | 218
score on a scale | 7.8 (4.8) | 7.6 (4.7)

ADVERSE EVENTS:
Time Frame: 1-month, 2-month, 4-month, 6-month
Description: No adverse effect is reported.
Arm/Group | Online Home-based Peer Support Intervention | Standard Usual Care
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/218
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/218
Other Adverse Events (participants affected / at risk) | 0/224 | 0/218

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT04621266/Prot_SAP_000.pdf